CLINICAL TRIAL: NCT06138704
Title: Retrograde Intrarenal Surgery Results and Stone-free Rate in Children With Kidney Stones
Brief Title: Evaluation of Retrograde Intrarenal Surgery Results and Stone-free Rate in Children With Kidney Stones
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Sponsor
Other Study IDs: E2-23-5305
Record Dates: First submitted 2023-11-14; First posted 2023-11-18 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Renal Stone; Retrograde Intrarenal Surgery
Keywords: Kidney Stone; Retrograde Intrarenal Surgery; Children; Stone Free Rate
MeSH Terms: conditions — Nephrolithiasis; Kidney Calculi

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Retrograde Intrarenal Surgery — All RIRS procedures were performed under general anesthesia with direct videoscopic and fluoroscopic guidance. The decision to use a flexible or semirigid ureteroscope depended on the location of the Stones. If this was not enough to pass the ureteroscope, we placed a JJ catheter for passive dilatation. Stones were fragmented using a holmium-YAG laser and grasped by a stone basket when applicable. Contrast injection was performed at the end of the procedures to confirm the absence of extravasation and stone-free status. Ultrasonography (USG) was performed three months, six months, and one year after the procedures to evaluate stone recurrence and hydronephrosis.
  Other Names: Lithohtrapsy

SUMMARY:
There is a global increase in the prevalence of urolithiasis in children attributed to lifestyle changes, dietary habits, climate changes, childhood obesity, and the wider availability of ultrasonography. The rising incidence of the disease with its recurrent nature emphasizes the need for minimally invasive therapeutic options. Patients in whom RIRS has been performed in the last four years with increasing experience will be presented, and complications, stone-free rates, and technical details will be discussed.

This retrospective Cohort study included children who underwent RIRS. Medical history, serum electrolytes, midstream urine culture, urinalysis, serum creatinine, complete blood count, and coagulation assessments were performed preoperatively. Ultrasonography (USG) was performed three months, 6 months, and 1 year after the procedures to evaluate stone recurrence and hydronephrosis. The investigators analyzed the stone-free rate ,complications, and the conversion to open procedure

DETAILED DESCRIPTION:
There has been a worldwide rise in the prevalence of urolithiasis in children, which is linked to changes in lifestyle and dietary habits, climate changes, childhood obesity, and the increased availability of ultrasonography (1). In pediatric stone disease, it is crucial to evaluate the underlying reasons, which may include metabolic disorders, anatomical anomalies, and infection, to avoid higher recurrence of stones after treatment (2). The increasing incidence and recurrence of this disease highlights the necessity for minimally invasive therapeutic solutions. Retrograde intrarenal surgery (RIRS) is gaining new indications owing to advanced laser and endoscopic technology, resulting in a constant rise in the number of procedures (3).

Routine RIRS has been performed in our clinic for the last 15 years with increasing rates. Patients in whom RIRS has been performed in the last three years with increasing experience will be presented, and complications, stone-free rates, and technical details will be discussed.

This retrospective cohort study included children who underwent RIRS between January 2019 and December 2022 at the Ankara Bilkent City Hospital, University of Health Science, Ankara, Turkey. The inclusion criteria were pediatric patients with kidney stones who underwent RIRS. The exclusion criteria were cases that were converted to open surgery, cases in which RIRS could not be performed because of anatomical reasons, and cases in which lower pole stones could not be reached with RIRS. The Ethics Committee of the Institution approved this study (E2-23-5305). All patient details were identified, and all patients provided written informed consent to participate in the study. Medical history, serum electrolytes, midstream urine culture, urinalysis, serum creatinine, complete blood count, and coagulation assessments were performed preoperatively. Plain abdominal film and ultrasonography/computer tomography scan examinations were also performed. Patients with preoperative positive urine culture results received a complete course of culture-specific antibiotics before RIRS Prophylactic antibiotic treatment with cephazolin was administered to all patients prior to surgery.

Surgical treatment was indicated when there was an obstruction, infection, failure of spontaneous stone passage, or stones larger than 7 mm and in the presence of increasing or unremitting colic.

All RIRS procedures were performed under general anesthesia with direct videoscopic and fluoroscopic guidance. All procedures were performed by the same surgeon. Semirigid ureteroscopy (4.5 Fr R. Wolf, Knittlingen, Germany) or flexible ureteroscopy (Karl Storz FLEX-X, Tuttlingen, Germany) was performed to place an access sheath. The decision to use a flexible or semirigid ureteroscope depended on the location of the stones. A flexible ureteroscope was used for lower pole stone, wherease a semirigid ureteroscope was preferred for renal pelvic or upper pole stones. In our practice, all children undergoing RIRS for stone disease received cephazolin. Perioperative antibiotic treatment was continued for a week following surgery. If a double J (JJ) stent was inserted, antibiotic prophylaxis was continued and ceased after removal of the JJ stent. A manual irrigation pump system was used for hydrodilation of the ureter during ureterorenoscopy. If this was not enough to pass the ureteroscope, the investigators placed a JJ catheter for passive dilatation. Ureteral active coaxial or balloon dilation was not performed. The investigators used isotonic fluid at body temperature to avoid hypothermia and hyponatremia during the procedures. The urinary bladder was maintained at low pressure with a 14-F suprapubic angiocatheter in all patients. Stones were fragmented using a holmium-YAG laser (Litho Quanta System, Italy) and grasped by a stone basket when applicable. Contrast injection was performed at the end of the procedures to confirm the absence of extravasation and stone-free status. The decision to place a postoperative uretral stent was made according to visible mucosal ureteral trauma or edema at the end of the procedure. The extracted stone specimens were submitted for stone analysis. All patients were discharged if fever was not detected the day after the procedures. Medical therapy and dietary planning were provided postoperatively on the basis of the composition of the stones. Ultrasonography (USG) was performed three months, six months, and one year after the procedures to evaluate stone recurrence and hydronephrosis. The investigators analyzed the stone-free rate, complications, and conversion to the open procedure. Statistical analysis was performed using the Chi-Square and ANOVA tests, p: 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria were pediatric patients with kidney stones who underwent RIRS.

Exclusion Criteria:

* The exclusion criteria were cases that were converted to open surgery, cases in which RIRS could not be performed because of anatomical reasons, and cases in which lower pole stones could not be reached with RIRS.

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: One hundred and five patients (49 boys and 56 girls) with a median age of 6,66+5,27 years (0,25-17,6 years) were treated with RIRS between January 2019 and December 2022. The RIRS procedure could not be performed in 15 cases, whereas it could be performed in 90 cases.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Determination of stone-free rate in children who underwent lithotripsy with retrograde intrarenal surgery for kidney stones. | USG evaluation was performed postoperative 1. month, 3-6-12-18 months, and kidney stones of the patients were evaluated.
  After the RIRS, patients were monitored with USG in the first month, 3-6-12 months, and stone-free rates were determined.

SECONDARY OUTCOMES:
How long does it take for renal stones to be cleared after RIRS? | USG evaluation was performed postoperative 1. month, 3-6-12-18 months, and kidney stones of the patients were evaluated.
  Patients first month after RIRS, 3-6-12. It was determined by follow-up with USG over the months and when stone-free status was achieved.
Determination of factors affecting stone-free rate in pediatric patients who underwent RIRS due to kidney stones. | USG evaluation was performed postoperative 1. month, 3-6-12-18 months, and kidney stones of the patients were evaluated.
  The effects of gender, age, number of stones, presence of staghorn stones, and whether a JJ stent was placed before the procedure on stone-free rates were evaluated in pediatric patients who underwent RIRS due to kidney stones.
Determining the need for repeated interventions to ensure stone-free status | Evaluating 4-year hospital records of patients
  The presence of additional interventions to ensure stone-free status was evaluated from hospital records.

OTHER OUTCOMES:
Determination of procedure-related complications in pediatric patients who underwent RIRS due to kidney stones. | Evaluating 4-year hospital records of patients
  Determination of procedure-related complications in pediatric patients who underwent RIRS due to kidney stones.

CONTACTS AND LOCATIONS:
Overall Officials: Huseyin T Tiryaki, MD, Study Director — University of Health Science Ankara Bilkent City Hospital
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Describe the IPD sharing plan, including what IPD are to be shared with other researchers.

REFERENCES:
- [Background] Clayton DB, Pope JC. The increasing pediatric stone disease problem. Ther Adv Urol. 2011 Feb;3(1):3-12. doi: 10.1177/1756287211400491. PMID 21789094
- [Background] Copelovitch L. Urolithiasis in children: medical approach. Pediatr Clin North Am. 2012 Aug;59(4):881-96. doi: 10.1016/j.pcl.2012.05.009. Epub 2012 Jun 15. PMID 22857835
- [Background] Azili MN, Ozcan F, Tiryaki T. Retrograde intrarenal surgery for the treatment of renal stones in children: factors influencing stone clearance and complications. J Pediatr Surg. 2014 Jul;49(7):1161-5. doi: 10.1016/j.jpedsurg.2013.12.023. Epub 2014 Jan 13. PMID 24952809
- [Result] Karagoz MA, Erihan IB, Doluoglu OG, Ugurlu C, Bagcioglu M, Uslu M, Sarica K. Efficacy and safety of fURS in stones larger than 20 mm: is it still the threshold? Cent European J Urol. 2020;73(1):49-54. doi: 10.5173/ceju.2020.0056. Epub 2020 Jan 3. PMID 32395324